CLINICAL TRIAL: NCT02064478
Title: Clinical Survey of Oticon Medical Ponto Implants and a Surgical Technique With Tissue Preservation
Status: Completed | Type: Observational
Sponsor: Oticon Medical (Industry)
Collaborators: Statistiska Konsultgruppen (Other)
Responsible Party: Sponsor
Other Study IDs: C47
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Conductive Hearing Loss; Mixed Hearing Loss; Single Sided Deafness
Keywords: Bone anchored hearing implant; Bone anchored hearing device
MeSH Terms: conditions — Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tissue preservation: Ponto implant installed using a tissue preservation surgical technique
- Tissue reduction: Ponto implant installed using a classical technique with skin thinning

SUMMARY:
A bone anchored hearing system is used to improve hearing for patients with e.g. conductive/mixed hearing loss or single sided deafness.

With this type of system, a titanium implant is installed in the temporal bone, where it osseointegrates, i.e. integrates with the bone. An abutment (also in titanium) is attached to the implants and penetrates the skin. The sound processor (hearing aid) is then connected to the abutment, and can be attached and removed by the patient via a snap-coupling. This type of system has been successfully implanted in more than 100.000 patients. Recently, a simplified surgical procedure, where no skin thinning around the abutment is made, was approved. The results after using this installation technique, here called soft tissue preservation, are the focus of this study.

The objective of the study is to compare the outcomes after a surgical procedure with soft tissue preservation (test) and a surgery with soft tissue reduction (control) for placing Oticon Medical Ponto implants and abutments. The main hypothesis is that patient numbness around the implant is less in the test group compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Patient indicated for an ear level bone anchored sound processor
* Bone thickness at the implant site of at least 4 mm

Exclusion Criteria:

* Inability to participate in follow-up
* Psychiatric disease in the medical history
* Mental disability
* Presumed doubt, for any reason, that the patient will be able to show up on all follow ups
* Diseases or treatments known to compromise the bone quality at the implant site, e.g. radiotherapy, osteoporosis, diabetes mellitus.
* Patients with natural skin height of >10 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients to be included are already planned for treatment with a bone anchored hearing aid at Radboud University Nijmegen Medical Centre (Nijmegen, The Netherlands).
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Numbness around implant, specifically mean Total sensibility | 36 months after surgery

SECONDARY OUTCOMES:
Length of surgery | At surgery
Sum of number of unplanned visits, revision surgeries, medications related to implant, and other treatments requiring medical staff per patient | 0-6 months
Mild/Adverse skin reaction | 0-6 months
  Adverse skin reaction is defined as a Holgers score ≥ 2 at least one follow-up visit, including unplanned visits, during the analysis period Holgers score is a standardized score of skin reactions around a bone anchored hearing implant.
Skin condition according to Holgers | 7 days after surgery
  Holgers score is a standardized score of skin reactions around a bone anchored hearing implant.
Postoperative complications | 7 days to 6 months
  Including
  * Bleeding or hematoma
  * Flap necrosis
  * Wound dehiscence
  * Other (description)
Proportion of patients with complete wound healing at first surgical visit | 7 days
Glasgow Benefit Inventory (GBI) scores | 3 months
Glasgow Health Status Inventory (GHSI) scores | Baseline (before surgery)
Abbreviated profile of hearing aid benefit (APHAB) scores | Baseline (before surgery)
Mean hours of use of the sound processor | 0-6 months
Sum of number of unplanned visits, revision surgeries, medications related to implant, and other treatments requiring medical staff per patient | 0-12 months
Sum of number of unplanned visits, revision surgeries, medications related to implant, and other treatments requiring medical staff per patient | 0-36 months
Bone conduction (BC) in-situ audiometric thresholds | 6 months
Bone conduction (BC) audiometric threshold | 6 months
  Measured with B-71
Mean total sensibility around implant | Baseline (before surgery)
Implant stability quotient (ISQ) | At surgery
Time to implant loss | 0-36 months
Patient and Observer scar assessment score | 21 days post surgery
Mild/Adverse skin reaction | 0-12 months
  Adverse skin reaction is defined as a Holgers score ≥ 2 at least one follow-up visit, including unplanned visits, during the analysis period
Mild/Adverse skin reaction | 0-36 months
  Adverse skin reaction is defined as a Holgers score ≥ 2 at least one follow-up visit, including unplanned visits, during the analysis period
Skin condition according to Holgers | 21 days
Skin condition according to Holgers | 12 weeks
Skin condition according to Holgers | 6 months
Skin condition according to Holgers | 1 year
Skin condition according to Holgers | 2 years
Skin condition according to Holgers | 3 years after surgery
Postoperative complications | 7 days to 12 months
  Including
  * Bleeding or hematoma
  * Flap necrosis
  * Wound dehiscence
  * Other (description)
Postoperative complications | 7 days to 36 months
  Including
  * Bleeding or hematoma
  * Flap necrosis
  * Wound dehiscence
  * Other (description)
Glasgow Benefit Inventory (GBI) scores | 12 months
Glasgow Health Status Inventory (GHSI) scores | 6 months
Glasgow Health Status Inventory (GHSI) scores | 36 months
Abbreviated profile of hearing aid benefit (APHAB) scores | 6 months
Abbreviated profile of hearing aid benefit (APHAB) scores | 36 months
Mean hours of use of the sound processor | 0-36 months
Mean total sensibility around implant | 21 days
Mean total sensibility around implant | 6 months
Mean total sensibility around implant | 12 months
Mean total sensibility around implant | 36 months
Implant stability quotient (ISQ) | 7 days post surgery
Implant stability quotient (ISQ) | 21 days post surgery
Implant stability quotient (ISQ) | 12 weeks post surgery
Implant stability quotient (ISQ) | 6 months post surgery
Implant stability quotient (ISQ) | 12 months post surgery
Implant stability quotient (ISQ) | 24 months post surgery
Implant stability quotient (ISQ) | 36 months post surgery
Patient and Observer scar assessment score | 6 months
Patient and Observer scar assessment score | 12 months
Patient and Observer scar assessment score | 36 months

OTHER OUTCOMES:
Skin height around abutment (in mm) | At surgery
Skin height around abutment (in mm) | 7 days post surgery
Skin height around abutment (in mm) | 21 days post surgery
Skin height around abutment (in mm) | 12 weeks post surgery
Skin height around abutment (in mm) | 6 months post surgery
Skin height around abutment (in mm) | 12 months post surgery
Skin height around abutment (in mm) | 36 months post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Myrthe KS Hol, MD, PhD, Principal Investigator — Radboud University Medical Center; Emmanuel AM Mylanus, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Centre, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] den Besten CA, Bosman AJ, Nelissen RC, Mylanus EA, Hol MK. Controlled Clinical Trial on Bone-anchored Hearing Implants and a Surgical Technique With Soft-tissue Preservation. Otol Neurotol. 2016 Jun;37(5):504-12. doi: 10.1097/MAO.0000000000000994. PMID 26945315